CLINICAL TRIAL: NCT03890029
Title: Building Biobehavioral Goal-Directed Resilience Among African American Women (Project GRIT)
Brief Title: G.R.I.T. - Goal-directed Resilience Intervention Training
Acronym: GRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Principal Investigator, Kisha Holden, PhD, MSCR, Professor, Morehouse School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1253996
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Chronic Post-Traumatic Stress Disorder
Keywords: PTSD; Elevated Cardiovascular Disease risk; Resilience
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Once potential participants have given consent and determined eligible, they will undergo an initial assessment.Pre, post- and follow-up testing. This consists of verbal scales including emotional well-being scales and mental health symptom scales. They will be administered in a group 30-60 minute session. Neuropsychological testing and psychophysiological tests given will require 90 minutes. Neuropsychological testing will be completed at pre and post testing only. In order to ensure unbiased assessment, pre- and post- and follow-up testing will be conducted by individuals blinded to study condition.
  Randomization. After pre-testing, all individuals will be randomly assigned to either the active treatment group or minimal attention control condition. After this, intervention participants will meet in small groups of 10 per group for 90 minutes/week over five weeks for resilience training. After five weeks, all participants will be post-tested.
  Interventions: Behavioral: Intervention Training
- Control (Other): While intervention participants receive resilience training, the control group will not receive training but will receive minimal attention of a bi-monthly telephone call to indicate to participants that they are still enrolled in the study. A monthly flyer will be mailed to them about wellness and PTSD in recent news coverage. Following completion of an intervention group, participants and controls will be scheduled for post-testing that will be identical to the pre-testing and will occur within two weeks after the final treatment session. After the post-testing and 3-month follow up testing, the controls will be offered the resilience training
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Intervention Training — After pre-testing and randomization, intervention participants will meet in small groups for 60 minutes/week over eight weeks for resilience training. Participants needing extra help will receive it at the end of each session. Controls will be on a minimal attention list, not being trained. After eight weeks, all participants will be post-tested.
  Arms: Intervention
Behavioral: Control Condition — While intervention participants receive resilience training, the control group will not receive training but will receive minimal attention of a bi-monthly telephone call to indicate to participants that they are still enrolled in the study. A monthly flyer will be mailed to them about wellness and PTSD in recent news coverage. Following completion of an intervention group, participants and controls will be scheduled for post-testing that will be identical to the pre-testing and will occur within two weeks after the final treatment session. After the post-testing and 3-month follow up testing, the controls will be offered the resilience training.
  Arms: Control

SUMMARY:
This research program has addressed three reactive adaptations evident in pain, PTSD, and obesity. In this project, the focus will be on PTSD as a model of stimulus-based reactive responses to unpredictability or threat, and the investigators propose to test the efficacy of the goal-directed skills training (GRIT) program for restoring predictive responding and homeostasis. The challenge of how best to cultivate psychological resilience in the face of stress, trauma, and social adversity among disadvantaged populations is a complex question best answered with a translational research approach. This research' intent is to help African American women who are dealing with stress after traumatic experiences. It will specifically study Post-traumatic Stress Disorder, a disorder that affects people who have experienced severe traumas. It is associated with a number of overwhelming emotional symptoms. These include sleep difficulties, depression and anxiety, flashbacks and nightmares of the traumatic events.

The training is an 8-week skill building program that helps people use positive experiences from their past to cope with current difficulties. The investigators will collect blood samples for future research to understand how the body's stress response changes as a result of this training

DETAILED DESCRIPTION:
This project will utilize an intervention that is to encompass tenets of the New Wave therapies in two important respects:

1. The project's emphasis is on capacity development. The project's focus reaches beyond symptoms to restore and build resilience strengths that nurture in the face of challenge. The concept of resilience first entered the psychological and psychiatric literature with the study of children suffering from stress and disadvantage who, nevertheless, were functioning well. Protective factors included the presence of caring adults and achievement at school . Bonds and achievement have remained the most persistent findings in decades of research .
2. The investigator's aim is to restore and build capacities displaced by symptoms. This will be accomplished by identifying the lost capabilities in narratives of survival and identifying neuroscience models that capture symptoms and lost capacities as bio-behavioral response systems that become visible in extreme environments. Narratives of exceptional survival in extreme situations are characterized by engagement with their circumstances in ways that kept individuals well, by social relatedness, and by an efficient stress response . For example, while imprisoned in the Hanoi Hilton, Robert Shumaker built a dream house and counted the feet of lumber and number of nails that would needed. Fellow inmates also developed a tapping code to communicate with each other. Thus, Shumaker was engaged, was socially connected through tapping and, while engaged, was not hyper-responsive to the threat around him. The positive survival responses are a marked contrast to the symptoms of PTSD described earlier, such as hyperarousal or intrusive thoughts. What distinguishes resilient adaptation in extreme situations from PTSD is that the resilient activities are characterized by goal-directed actions while PTSD is characterized by stimulus-driven responses. The distinction of goal-directed versus stimulus-based responding is extensively developed in the neuroscience and cognitive literature. Action research has identified intention-based and stimulus-based actions in which self-initiated actions involve brain mechanisms and cognitive processes distinctly different from reflexive or responsive movement.

Broadly conceived, humans have two types of responses to the environment: they act to achieve results or goals in the environment, thus changing the environment, or they respond to and accommodate the demands of the environment and are changed by it. This distinction has its parallels in other areas of human functions. Attention studies have identified voluntary control of attention (endogenous) that is goal-directed versus automatic reflexive control (exogenous) in which external objects or events claim a subject's attention. A number of cortical models are relevant to goal-directed action and stimulus-based responding, among them the work on intention and reactivity by Astor-Jack and Haggard or the studies of Hannus and colleagues on stimulus-driven and user-driven control of visual attention.

Perhaps most relevant is the predictive and reactive control system (PARCS) developed by Tops and colleagues.

These two basic bio-behavioral programs control behavior in different environments, the reactive program being most adaptive in unpredictable environments and the predictive program most effective in highly predictable environments. The reactive program is guided by momentary feedback from the environment and responses are close in time and space. The predictive program guides behavior in a feed-forward manner that plans for the future, simulates alternatives, and makes predictions. In PTSD, stimulus-based responding prevails and displaces goal-directed responding at multiple levels of functioning: cortical, endocrine, affective, cognitive - indeed, the entire bio-behavioral system of predictive responding.

The abundant research on goal-directed action versus stimulus-based responding has few parallels in clinical psychology or psychiatry. Hints emerge in eudamonic well-being that is goal-directed and required for challenging situations and goal-relevant motivational constructs of self-efficacy or locus of control. This study draws on the extensive neuroscience framework to formulate a model of resilient and traumatic responses and proposes an approach that restores goal-directed responding that will simultaneously reduce the dominance of stimulus based symptoms of PTSD. This is a 5 year study with the anticipation of 148 enrolled.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black (self-identified)
* Diagnosis of PTSD
* Between the ages of 18-64 other illnesses due to aging, cognitive declines due to aging, retirement change in life demands at age 65.
* Able and willing to provide consent

Exclusion Criteria:

* Active suicidality
* Active alcohol and substance use of moderate or severe levels of severity
* Psychosis
* Current severe disabling illness (recent surgery, impending surgery, extreme pain interfering with participation)
* Unable to meet attendance requirements: limit of 2 missed session of the 8.
* Not engaged in other therapies for PTSD, cognitive behavior therapy, exposure therapy and reprocessing therapy.
* Unable to participate in small group interactive setting.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Clinician Administered PTSD Scale for DSM 5 (CAPS-5): clinician-administered, structured interview ideal for screening, differential diagnosis & confirmation of PTSD. Each item is scored on a scale of 0-4; the total composite score range is 0-212; Lower score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the PTSD Checklist (PCL-5): 17-item self-report checklist of PTSD symptoms; General civilian version of the PCL will be used. Each item is scored on a scale of 0-4; the total composite score range is 0-80; Lower score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Posttraumatic Cognitions Inventory (PTCI): 36-item self-report measure assessing trauma-related thoughts and beliefs about self, others, and self-blame. Each item is scored on a scale of 1-7; the total composite score range is 33-231; Lower score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Difficulties in Emotion Regulation: 36-item self-report questionnaire designed to assess multiple aspects of emotion dysregulation. Each item is scored on a scale of 1-5; the total composite score range is 36-180; Lower score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Positive & Negative Affective Schedule (PANAS): 20-item self-report measure frequently used as a measure of general affective states. Each item is scored on a scale of 1-5; the total composite score range is 20-100; 1=very slightly or not at all; 5=extremely; measures positive and negative affect mood scales; higher scores on positive affective scale and lower scores on negative affective scale indicate better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Ryff Scales of Psychological Well-being: Measures aspects of psychological well-being across three selected subscales: Personal Growth, Positive Relations with Others, Purpose in Life; 9 items each. Each item is scored on a scale of 1-7; the total composite score range is 7-42; Higher score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Conner-Davidson Resilience Scale (CD-RISC): Unidimensional self-reported scale consisting of 10 items measuring resilience. Each item is scored on a scale of 0-4; the total composite score range is 0-100; Higher score = better outcome
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): Originally designed to identify and characterize mild and severe dementia in older adults, later modified to include younger adults. This study will focus on immediate memory, delayed memory, simple and complex attention subtests. In the Immediate memory subset the participant is asked to recall words from a list immediately after being read to her/him; More words remembered = better outcome. In the Delayed memory subset the participant asked to recall words from a list some time after being read to her/him; More words remembered = better outcome, In the Simple attention subset the participant is asked to repeat increasingly longer sequences of digits; More/longer sequences remembered = better outcome. In the Complex attention subset the participant matches symbols with numbers; More correct matches = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Delis-Kaplan Executive Function System (D-KEFS): Study focuses on two of nine subtests (Verbal Fluency and Color-Word Interference) assessing components of executive functioning. In the Verbal Fluency subset the participant says words that begin with a specified letter, belong to a designated semantic category, and alternate between saying words from two different semantic categories; More words participant can say per category = better outcome. In the Color-Word Interference subset the participant names color patches, reads words naming colors printed in black ink, names the ink color in which color words are printed in an incompatible ink color, and switches back and forth between naming the dissonant ink color and reading the conflicting words; More accurate = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by demographics: Collected demographic data will include age, gender, race, etc. Each item is scored on a scale of 0-3; the total composite score range is 0-66; Lower score=better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Beck Depression Inventory (BDI): reflects DSM criteria for depression, score indicates presence of minimal, mild, moderate, or severe depressive symptoms. Each item is scored on a scale of 0-3; the total composite score range is 0-66; Lower score=better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Patient Health Questionnaire Depression Scale (PHQ-9): 9-item measure reflecting DSM criteria for depression. Each item is scored on a scale of 0-3; the total composite score range is 0-27; Lower score = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Alcohol Use Disorders Identification Test (AUDIT-C): brief alcohol screen used to identify persons who have active alcohol use disorders, including alcohol abuse or dependence. Each item is scored on a scale of 0-4; the total composite score range is 0-68; For each item, a score of 4 or more in men and 3 or more in women is considered positive, optimal for identifying hazardous drinking or active alcohol use disorders; Lower score = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the SF-36 Health Measures: Multi-purpose, short-form health questionnaire of functional health and well-being scores. Over seven subsections, seven items are scored on a scale of 1-2 for a total composite score range of 7-14; ten items are scored on a scale of 1-3 for a total composite score range of 10-30; nine items are scored on a scale of 1-5 for a total composite score range of 9-45; and ten items are scored on a scale of 1-6 for a total composite score range of 10-60; Lower score = better outcome for 16 items; Higher score = better outcome for 20 items.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Mini International Neuropsychiatric Interview (MINI): Short diagnostic structured interview designed to assess various psychiatric disorders according to DSM-IV and ICD-10 criteria. 98 items on a Yes/No scale with a skip pattern (i.e. not all 98 questions will necessarily be answered) and 49 qualitative questions; Fewer reported symptoms = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Berlin Questionnaire: self-reported questionnaire assessing snoring, sleepiness or fatigue, obesity and hypertension. Ten questions over three categories with non-uniform, symptom specific self-ratings; Positive (worse outcome) ranges are color-coded on the questionnaire.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Pittsburgh Sleep Quality Index (PSQI): self-rated questionnaire that assesses sleep quality, latency, duration, efficiency, disturbances, sleep medication, and daytime dysfunction over a one-month time interval. Six qualitative questions, 17 questions rating symptoms from "Not during the past month" to "Three or more times a week"; More answers of "Not during the past month" = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Epworth Sleepiness Scale (ESS): self-report instrument on which respondents rate their chance of falling asleep in eight common daily situations. Each item is scored on a scale of 0-3; the total composite score range is 0-24; Lower score = better outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Short Form McGill Pain Questionnaire (SF-MPQ): 15 descriptors (11 sensory, 4 affective) rated on intensity scale (1=mild, 2=moderate, 3=severe, 4=none) the total composite symptomatic score range is 15-45; Lower symptomatic score = better outcome; 60 (no symptoms on any of the items)=best outcome.
Effects of a resilience building intervention on psychological, cardiovascular risk and resilience outcomes in a group of African American women with clinically significant posttraumatic stress symptoms | 3-6 months
  Changes in pre-to-post scores among intervention versus control group as measured by the Structured Trauma Interview (STI): A non-invasive test that gathers specific information about trauma-related cognitive and physiological symptoms. A clinician administers qualitative questions to participants hooked up to machines that record physiological reactions (e.g. heart rate); Lower physiological response=better outcome.

SECONDARY OUTCOMES:
Effects of fear, cardiovascular physiology, and sleep patterns on response to a resilience building intervention in a group of African American women with clinically significant posttraumatic stress symptoms | 12 months
  Changes in pre-to-post measures among intervention versus control group as assessed by Actigraphy, a non-invasive approach to monitoring sleep/activity cycles that will collect five days of sleep data to assess sleep/wake behavior, circadian rhythm, and effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kisha B Holden, PhD, MSCR, Principal Investigator — Morehouse School of Medicine
Locations (2):
- United States (2):
  - Grady Health Systems, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research project will utilize the Morehouse School of Medicine Community Engagement Core for local, regional and national dissemination of findings. A community-based knowledge exchange event will be conducted in 3-5 years
Time Frame: 3-5 years